CLINICAL TRIAL: NCT05991024
Title: Pulmonary Ventilation Function Between Patients With Primary and Recurrent Incisional Hernia: a Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Director, Fudan University
Other Study IDs: HuadongHosptialHernia
Record Dates: First submitted 2023-08-05; First posted 2023-08-14 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Incisional Hernia; Recurrent Hernia; COPD; Pulmonary Ventilation Function
Keywords: Incisional Hernia; Recurrent Hernia; COPD; Pulmonary ventilation function
MeSH Terms: conditions — Incisional Hernia; Hernia; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The primary group: Patients diagnosed with "incisional hernia" in our hospital's electronic medical record system were divided into two groups: primary group and recurrent group based on whether the incisional hernia recurred after incisional hernia repair,who were screened out with abdominal wall incisional hernia.
- The recurrent group: Patients diagnosed with "incisional hernia" in our hospital's electronic medical record system were divided into two groups: primary group and recurrent group based on whether the incisional hernia recurred after incisional hernia repair,who were screened out with abdominal wall incisional hernia.
  Interventions: Behavioral: the incisional hernia recurrent

INTERVENTIONS:
Behavioral: the incisional hernia recurrent — Recurrence after repair was the main outcome
  Groups: The recurrent group

SUMMARY:
Purpose Chronic obstructive pulmonary disease (COPD) is a risk factor for incisional hernia, COPD has persistent airflow restriction and pulmonary ventilation dysfunction. The aim of this study was to compare differences in pulmonary ventilation function between primary incisional hernia and recurrent incisional hernia.

Method According to the inclusion and exclusion criteria,Patients diagnosed with "incisional hernia" in our hospital's electronic medical record system were divided into two groups: primary group and recurrent group based on whether the incisional hernia recurred after incisional hernia repair,who were screened out with abdominal wall incisional hernia.The patient information of the two groups were collected, examined and recorded.The clinical data was analyzed by using statistical analysis software.

DETAILED DESCRIPTION:
Method Study design and patient population： This study is a single-center cross-sectional study. The main steps of this study are patients search, information review, data record, data verification and statistical analysis.

The investigators searched the electronic medical record system from January 2016 to March 2023, using the 10th edition of the International Classification of Diseases (ICD-10).

Inclusion and exclusion criteria The investigators reviewed the physical examination records of each patient, combined with abdominal CT images, only patients diagnosed with "abdominal incisional hernia" were included in our study, patients with other types of abdominal external hernia, such as parastomal hernias and umbilical hernias, were excluded.

CT imagings of the abdomen and pulmonary function tests were two required items. Patients with incomplete data were excluded, patients with complete data were included in the study and were divided into two groups: primary group and recurrent group depends on whether there is a recurrence.

Because primary incisional hernia may turn into recurrence. To reduce error, patients with primary incisional hernia less than one year when the study was started were excluded, the investigators conducted telephone follow-up of patients with primary incisional hernia. Recurrence after repair was the main outcome, patients with follow-up results of non-recurrence were included in the study. Patients who have recurrent require reassessment of pulmonary function, the patients with missing pulmonary function are excluded.

The search was carried out by two researchers who extracted data independently and the results were double-checked; Diagnosis is done independently by two experienced surgeons, based on medical history and CT images. If there is disagreement, it will be determined after discussion with a third experienced surgeon.

Data Collection The investigators extracted the patient's age, gender, ethnicity, BMI, abdominal CT image, maximum length of abdominal wall defect, hypertension, diabetes, coronary heart disease and pulmonary function test report, pulmonary function test including pulmonary ventilation function and pulmonary diffusion function, pulmonary ventilation function is the main observation index of this study. The fixed threshold method often used in China to grade pulmonary ventilation dysfunction[9], our hospital graded the severity of pulmonary ventilation dysfunction with FEV1 as a percentage of the expected value: Mild: >70%; Moderate: 60%~69%; Moderate to severe: 50%~59%; Severe: 35%~49%; Very severe: <35%. The maximum length of the abdominal wall defect is measured using multi-slice helical CT 3D reconstruction technology, which is performed by a radiologist.

Statistical analysis Continuous variables that conform to a normal distribution are tested using an independent sample t-test; Chi-square test and continuous correction chi-square test are used for categorical variables; The grading variables use Wilcoxon's sum test. When P<0.05, the difference was considered statistically significant, and the statistical analysis software used in this study was SPSS Version 20.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal incisional hernia
* Complete CT imagings of the abdomen and pulmonary function tests data

Exclusion Criteria:

* Abdominal external hernia, such as parastomal hernias and umbilical hernias
* Primary incisional hernia less than one year when the study started

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed with "abdominal incisional hernia"and complete data
Sampling Method: Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Recurrent | 2016.1-2023.3
  Recurrence after surgery repair

CONTACTS AND LOCATIONS:
Locations (1):
- Yiming Lin, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
I have to make sure that the patient's privacy and rights are adequately protected